CLINICAL TRIAL: NCT01409863
Title: A Comparison Evaluation of Fractional Laser Therapy an Dermabrasion for Scar Revision
Brief Title: Fractional Laser Therapy and Dermabrasion for Scar Revision
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has left University of Minnesota.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1001M75732
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Scar
Keywords: post surgical or post traumatic scar on face or scalp
MeSH Terms: conditions — Cicatrix | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- laser and standard diamond fraise dermabrasion (No Intervention): laser and standard diamond fraise dermabrasion
  Interventions: Procedure: laser and standard diamond fraise dermabrasion

INTERVENTIONS:
Procedure: laser and standard diamond fraise dermabrasion — standard dermabrasion, CO2 laser resurfacing

SUMMARY:
The goals of this study will be to compare the safety and efficacy of fractional photothermolysis (Fraxel) with dermabrasion when used for scar revision.

DETAILED DESCRIPTION:
Post traumatic and post surgical scar resurfacing is a common reason for patient visits to dermatologists and plastic surgeons. The Fraxel Laser is a new FDA cleared treatment for textural irregularities of the skin. There have been no studies examining the efficacy of Fraxel specifically for scar resurfacing though it is being used in clinical practice as its clearance was given under hte umbrella of "coagulation of soft tissue." Dermabrasion is the gold standard for scar resurfacing and provides the criterion against which Fraxel therapy should be measured.

ELIGIBILITY:
Inclusion Criteria:

* post surgical or post traumatic scar on face or scalp
* age 18 or older
* able to read and comprehend English
* Willing to follow treatment schedule and post treatment care requirements
* signed informed consent form
* Fitzpatrick skin type I-III

Exclusion Criteria:

* known photosensitivity
* taken any medications known to induce photosensitivity in previous three months
* taken accutane within past 12 months
* pregnant or nursing
* currently on topical or oral antibiotics
* immunocompromised status
* skin type IV or greater

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
safety and efficacy of fractional photothermolysis | Post Surgery
  compare the safety and efficacy of fractional photothermolysis (Fraxel) with dermabrasion when used for scar revision.

CONTACTS AND LOCATIONS:
Overall Officials: John Christophel, MD, Principal Investigator — University of Minnesota